CLINICAL TRIAL: NCT01386255
Title: Placebo Controlled Study of Baclofen for GERD in Children With Cerebral Palsy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants were enrolled
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Samuel Nurko, Attending Physician; Director, Center for Motility and Functional Gastrointestinal Disorders, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Baclofen-07-02-0077; 1R21DK077678-01 (NIH)
Record Dates: First submitted 2011-06-29; First posted 2011-07-01 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Cerebral Palsy; GERD
Keywords: GERD
MeSH Terms: conditions — Cerebral Palsy; Gastroesophageal Reflux | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- baclofen (Active Comparator): Baclofen suspension
  Interventions: Drug: Baclofen
- placebo (Placebo Comparator): Identical palcebo suspension
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Baclofen — The final baclofen dose will be 0.7 mg/kg (to a maximum of 40 mg/day) divided in three doses.
  Other Names: Lioresal
  Arms: baclofen
Drug: placebo — placebo. No other names
  Arms: placebo

SUMMARY:
Despite the use of proton pump inhibitors and available prokinetics, medical therapy is ineffective in an important number of children with cerbreal palsy (CP) and gastroesophageal reflux disease (GERD), and failure of medical therapy is associated with a substantial morbidity. Many patients, particularly children with CP and GERD, continue to experience complications despite aggressive therapy because antisecretory medications do not address the primary reflux mechanism (TLESR). Furthermore, in patients with CP, surgical options are fraught with serious complications and long-term morbidity. Because the available treatment options for children with CP and intractable GERD are limited, new therapies are urgently needed. Baclofen, which has been shown in animals and humans to decrease TLESRs, may be a good alternative for the treatment of children with CP with intractable GERD.

DETAILED DESCRIPTION:
Despite the use of proton pump inhibitors and available prokinetics, medical therapy is ineffective in an important number of children with cerbreal palsy (CP) and gastroesophageal reflux disease (GERD), and failure of medical therapy is associated with a substantial morbidity. Many patients, particularly children with CP and GERD, continue to experience complications despite aggressive therapy because antisecretory medications do not address the primary reflux mechanism (TLESR).

This is a placebo controlled trial of baclofen for the treatment of GERD in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* 3-18 years old
* Diagnosis of Cerebral Palsy
* Symptoms of GERD for at least 3 months
* At least 8 weeks on BID therapy with a PPI at a therapeutic dose at time of enrollment
* Normal upper gastrointestinal barium contrast study (UGI)
* Have a g-tube that is used for more than 75% of calories and a stable feeding schedule for at least 2 weeks
* If seizures are present, they need to be controlled and on stable medications for 4 weeks

Exclusion Criteria:

* Underlying electrolyte disturbance
* History of Nissen fundoplication
* Renal insufficiency
* Currently receiving baclofen
* Baclofen allergy
* Uncontrolled seizure disorder
* Lack of informed consent

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04-30 (Actual)

PRIMARY OUTCOMES:
Symptom control | 3 weeks
  Symptom frequency during the 2 weeks of placebo and baclofen administration.

SECONDARY OUTCOMES:
GERD control | 3 weeks
  Frequency and duration of reflux episodes detected by MII during 24 hours of recording after two weeks of maximum dose.
  Proportion of full-column and non-acid reflux episodes detected by MII during 24 hours after two weeks of maximum dose.
  Frequency of TLESRs and reflux associated with TLESRs at half of the maximum dose, and after two weeks of maximum dose are administered
side effects of baclofen | 3 weeks
  Incidence of side effects and rate of discontinuation of the study

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Nurko, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States